CLINICAL TRIAL: NCT01656447
Title: The Scleroderma Registry & Repository
Brief Title: Scleroderma Registry & Repository at the Hospital for Special Surgery
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-276
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Scleroderma
Keywords: Scleroderma; Scleroderma Registry; Hospital for Special Surgery Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Research bloods will be collected if the patient gives permission. These bloods can be donated at the time of a patient's private visit with a physician at Hospital for Special Surgery, or at an independent research visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Scleroderma: Patients who have been diagnosed at any point in their life with Scleroderma will compose the cohort.

SUMMARY:
The overall objective of the Scleroderma Registry is to support and promote the basic science and clinical research of this complex rheumatic disease at the Hospital for Special Surgery (HSS). The registry facilitates our understanding of the clinical features, pathobiology, genetics of Scleroderma. This will ultimately lead to a potential treatment for this currently untreatable condition.

DETAILED DESCRIPTION:
What will be asked of you:

* Completion of 2 health questionnaires
* Donation of research bloods. This is optional, but encouraged (if possible).
* We also encourage patients who come for initial visits to return so follow-up data can be collected.

Benefits to Patients:

* The HSS Scleroderma Registry gives patients the opportunity to participate in observational research with the goal of improving the lives of patients in the future.
* By donating research bloods and providing clinical information, patients will help generate new knowledge about Scleroderma that can guide the treatment and care of patients afflicted with this rare disease.
* Patients will also receive a comprehensive, medical evaluation from an HSS physician who specializes in treating Scleroderma. He or she will provide guidance on treatment options and recommendations for current or upcoming clinical trials.
* Physicians will also make patients aware of the resources available to them, including support groups and educational programs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals older than 18 years of age with Scleroderma

Exclusion Criteria:

* Individuals younger than 18 years of age
* Individuals older than 18 years of age without Scleroderma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individuals older than 18 years of age who have Scleroderma
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-08; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rodnan Skin Score | Baseline & follow-up visits during regularly scheduled appointments for up to 5 years
  Physician score of skin thickening over 17 areas of the body.

SECONDARY OUTCOMES:
Scleroderma Health Assessment Questionnaire | Baseline & follow-up visits during regularly scheduled appointments for up to 5 years
  Patient questionnaire
Short Form-36 | Baseline & follow-up visits during regularly scheduled appointments for up to 5 years
  Patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Spiera, MD, Principal Investigator — Hospital for Special Surgery, New York; Jessica K Gordon, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- See also: Scleroderma, Vasculitis, & Myositis Center Website — http://www.hss.edu/scleroderma-vasculitis-center.asp